CLINICAL TRIAL: NCT02322905
Title: Cancer Caregiver Burden: Targeting Emotion Regulation in a Randomized Controlled Trial
Brief Title: Cancer Caregiver Burden: Targeting Emotion Regulation in a Trial
Acronym: ERT-ICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ERT15-17
Record Dates: First submitted 2014-12-04; First posted 2014-12-23 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Depression
Keywords: informal caregivers; caregiving; psychotherapy for caregivers; cancer; emotion regulation; distress; inflammation
MeSH Terms: conditions — Neoplasms; Emotional Regulation; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emotion Regulation Therapy (Experimental): 8 sessions of Emotion Regulation Therapy.
  Interventions: Behavioral: Emotion Regulation Therapy
- Usual Medical Care (No Intervention): No planned psychotherapy.

INTERVENTIONS:
Behavioral: Emotion Regulation Therapy — 8 sessions of ERT
  Arms: Emotion Regulation Therapy

SUMMARY:
Informal caregivers of cancer patients report high levels of psychological distress as evidenced in markedly increased levels of anxiety and depression. High levels of psychological distress in caregivers have also been found to be associated with poorer health and increased levels of pro-inflammatory cytokines that are well-established risk factors for physical illness and stress-related mortality. Previous psychological interventions using cognitive methods have only produced small effect sizes and more research on how to effectively alleviate caregiver burden is needed. The proposed project will investigate the effect of Emotion Regulation Therapy (ERT) for caregivers of cancer patients. ERT is a novel approach specifically targeting emotion regulation with the aim of improving mental and physical health. The effect of ERT will be examined in a randomized controlled trial comparing ERT to usual medical care (UMC).

DETAILED DESCRIPTION:
PURPOSE:

The primary purpose of the study is to test the efficacy of Emotion Regulation Therapy (ERT) for informal caregivers (ICs) of cancer patients. ERT is a manualized treatment for ICs and consists of 8 weekly sessions.

AIMS AND HYPOTHESES:

Intervention and mediation effects. In an RCT, the investigators will investigate the efficacy of an 8 session ERT for ICs on psychological and physical distress and a number of other health outcomes in both ICs and cancer patients. Outcomes in the ERT group will be compared to outcomes in a group of ICs and patients receiving usual medical care (UMC) (see Figure 1). ICs receiving ERT compared to ICs receiving UMC are expected to exhibit 1a) significant reductions in psychological distress and perceived caregiving burden, 1b) improvements in quality of life; and 1c) improvements in pro-inflammatory markers of stress/immune functioning. Likewise, patients whose ICs receive ERT are expected to report 2a) reduced anxiety and depression, 2b) improved quality of life and 2c) less chronic inflammation. Due to the design, these effects will be considered following the acute treatment period (pre, mid and post therapy). In addition to this, gains are expected to be maintained over the follow-up-period. In addition, 3) improvements are exptected to be maintained over the follow-up period. Finally, 4) improvements in adaptive emotion regulation (mindfulness, acceptance, and cognitive reappraisal) are expected to mediate the effect of ERT.

PARTICIPANTS AND PROCEDURES:

ICs of cancer patients with various cancer types will be consecutively recruited from Aarhus University Hospital, Denmark. Staff at the Outpatient Clinic at the Department of Oncology, Aarhus University Hospital, Denmark, will screen ICs at the department. Initially the investigators wanted to include caregivers of patients with lung and colorectal cancer only. However, in order to be able to include caregivers at a faster pace, it was decided - after one month during which only two caregivers were included - to broaden the patient group. Furthermore, it was decided that more than one IC per patient could participate.

After giving informed consent, participants will be randomized to Emotion Regulation Therapy (ERT) or usual medical care (UMC) in a ratio of 1:1 by means of computer-generated randomization lists. Outcome measures will be obtained pre-, mid-, and post-therapy as well as at 3 and 6-month follow-up. At every ERT session, ICs and clinicians will fill out a number of self-report the process measures. Cancer patients will be assessed pre- and post ERT, and at 3 and 6-months follow-up. Every IC and patient will provide blood samples before and after the intervention as well as at follow-ups.

Based on a power calculation (alpha=0.0125, beta=0.90), a dropout rate of 35%, and an intraclass correlation between ICs of the same patient of 0.20, the inclusion of 80 ICs will allow for an interaction effect between group (ERT vs. UMC) and time (acute treatment, thats is, pre, mid and post) of a medium effect size (d=0.5) to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Medium levels of distress (distress thermometer > 3) and at least moderate levels of worry or rumination
* Caregiver of patient with cancer

Exclusion Criteria:

* an expected survival of the patient of <6 months,
* active substance abuse (alcohol or drugs), and
* participation in other psychosocial trials.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in The Caregiver Reaction Assessment and EORTC-QLQ-30 | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring burden in ICs and quality of life cancer patients, respectively
Change in Hospital Anxiety and Depression Scale (HADS) | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring anxiety and depression
Change in Penn State Worry Questionnaire | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring worry
Change in Rumination Response Scale - Brooding subscale only | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring brooding

SECONDARY OUTCOMES:
Change in Difficulty in Emotion Regulation Scale | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring emotion regulation
Change in Emotion Regulation Questionnaire | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring emotion regulation
Change in Five Facet Mindfulness Questionnaire | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring mindfulness
Change in Experiences Questionnaire | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring psychological distancing
Change in The Pittsburgh Sleep Quality Index | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring sleep quality
Change in quality of life - WHO-5 | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring quality of life
Change in Pro-inflammatory markers: CRP, TNFalpha, IL-1, IL-6 | Between-group effect at post, based on the whole treatment duration (pre-, and post-therapy).
  Serum-derived pro-inflammatory markers (only pre and post therapy)
Emotional closeness | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  2 items (actual and wanted emotional closeness) rated on a 0-10 scale
Emotional attention coping (EAC) | Between-group effect at post, based on the whole treatment duration (pre-, mid- and post-therapy).
  Questionnaire measuring emotion regulation

CONTACTS AND LOCATIONS:
Overall Officials: Mia S O'Toole, MSc, Principal Investigator — University of Aarhus
Locations (1):
- Unit for Psychooncology and Health Psychology, Aarhus C, Denmark

REFERENCES:
- [Derived] Mikkelsen MB, Elkjaer E, Mennin DS, Fresco DM, Zachariae R, Applebaum A, O'Toole MS. The impact of emotion regulation therapy on emotion differentiation in psychologically distressed caregivers of cancer patients. Anxiety Stress Coping. 2021 Jul;34(4):479-485. doi: 10.1080/10615806.2021.1929934. Epub 2021 May 28. PMID 34047220